CLINICAL TRIAL: NCT01306786
Title: Five Days Quadruple and Clarithromycin Containing Triple Therapy as Empirical First and Second-Line Treatment for Helicobacter Pylori Eradication: a Randomized Crossover Trial
Brief Title: Five Days Quadruple and Clarithromycin Containing Triple Therapy as Treatment for Helicobacter Pylori Eradication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr Ivan FN Hung, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HKU-HP1
Record Dates: First submitted 2011-02-24; First posted 2011-03-02 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Helicobacter Pylori Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quadruple therapy (Active Comparator): First line: 5 days esomeprazole 20mg b.d., bismuth subcitrate 120mg q.i.d., tetracycline 250mg q.i.d. and metronidazole 250mg q.i.d.
  Cross over second line for those who failed first line: 7 days esomeprazole 20mg b.d., amoxicillin 1g b.d. and clarithromycin 500mg b.d
  Interventions: Drug: Quadruple therapy
- Triple Therapy (Active Comparator): First line: 7 days esomeprazole 20mg b.d., amoxicillin 1g b.d. and clarithromycin 500mg b.d Second line cross over if failed first line: 7 days quadruple therapy: esomeprazole 20mg b.d., bismuth subcitrate 120mg q.i.d., tetracycline 250mg q.i.d. and metronidazole 250mg q.i.d.)
  Interventions: Drug: Triple therapy

INTERVENTIONS:
Drug: Quadruple therapy — First line: 5 days esomeprazole 20mg b.d., bismuth subcitrate 120mg q.i.d., tetracycline 250mg q.i.d. and metronidazole 250mg q.i.d.
  Cross over second line for those who failed first line: 7 days esomeprazole 20mg b.d., amoxicillin 1g b.d. and clarithromycin 500mg b.d
  Arms: Quadruple therapy
Drug: Triple therapy — First line: 7 days esomeprazole 20mg b.d., amoxicillin 1g b.d. and clarithromycin 500mg b.d Second line cross over if failed first line: 7 days quadruple therapy: esomeprazole 20mg b.d., bismuth subcitrate 120mg q.i.d., tetracycline 250mg q.i.d. and metronidazole 250mg q.i.d.)
  Arms: Triple Therapy

SUMMARY:
The aim of this randomized trial is to compare the efficacy and tolerability of H. pylori eradication with a 5-day quadruple therapy versus a clarithromycin-containing triple therapy.

DETAILED DESCRIPTION:
Eligible patients with H pylori infection were randomized to receive either five-day QUAD (esomeprazole 20mg b.d., bismuth subcitrate 120mg q.i.d., tetracycline 250mg q.i.d. and metronidazole 250mg q.i.d.) or EAC (esomeprazole 20mg b.d., amoxicillin 1g b.d. and clarithromycin 500mg b.d.). H. pylori status was rechecked by 13C urea breath test 8 weeks after treatment. Patients who failed their respective therapy were invited to undergo H. pylori susceptibility testing and crossover to receive the alternative regimen for the same duration.

ELIGIBILITY:
Inclusion Criteria:

* patients with H. pylori infection
* did not receive H. pylori eradication therapy before

Exclusion Criteria:

* patients who have received previous H. pylori eradication therapy
* co-morbidity of liver cirrhosis
* co-morbidity of renal failure
* co-morbidity of alcoholism
* co-morbidity of malignancy
* received antibiotics, bismuth preparations, proton pump inhibitors or probiotic in the preceding three months
* patients with known allergy to the medications used
* patients with a history of previous gastrointestinal diseases or gastric surgery
* pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
H pylori eradication | 8 weeks after treatment
  Successful H pylori eradication documented by urea breath test after first and second line treatments. Cross over if patients failed first line treatment

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 10 weeks outpatient follow-up
  Assessed adverse effects and compliance by standard questionnaire upon 10 weeks outpatient follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ivan F Hung, MD MRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong SAR, Hong Kong